CLINICAL TRIAL: NCT05603884
Title: Venetoclax Combining Chidamide and Azacitidine (VCA) Regimen Followed by Dicitabine Combined With Liposome Mitoxantrone, Cytarabine, and G-CSF (D-MAG) Regimen on the Treatment of Elderly Patients With Newly Diagnosed Acute Myeloid Leukemia (AML) : A Multicenter, Prospective, Single Arm Clinical Trial
Brief Title: VCA Regimen Followed by D-MAG Regimen on the Treatment of Elderly Patients With Newly Diagnosed Acute Myeloid Leukemia (AML)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Collaborators: Chipscreen Biosciences, Ltd. (Industry); CSPC Pharmaceutical Group Limited (Industry); Fujian Provincial Hospital (Other); Fujian Cancer Hospital (Other Government); Zhangzhou manicipal hospital of Fujian Province (Unknown); Jieyang People's Hospital (Other); Huizhou Municipal Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FXMH-AML-002; ChiCTR2200061925 (Registry Identifier: Chinese clinical trial registry)
Record Dates: First submitted 2022-10-29; First posted 2022-11-03 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Leukemia, Myeloid, Acute; AML Stage, Adult
Keywords: newly diagnosed acute myeloid leukemia; liposome mitoxantrone; sequential treatment
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Azacitidine; Cytarabine; Granulocyte Colony-Stimulating Factor; Clinical Protocols

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment arm (Experimental): 2 cycles of VCA regimens followed by 2 cycles of D-MAG regimens, and then repeat the above four courses of treatment once
  Interventions: Drug: Venetoclax Combining Chidamide and Azacitidine (VCA) regimen followed by dicitabine combined with liposome mitoxantrone, cytarabine, and G-CSF (D-MAG) regimen

INTERVENTIONS:
Drug: Venetoclax Combining Chidamide and Azacitidine (VCA) regimen followed by dicitabine combined with liposome mitoxantrone, cytarabine, and G-CSF (D-MAG) regimen — venetoclax combining chidamide and azacitidine (VCA) 28 days per cycle × 2 cycles； 1) chidamide 30mg biw × 2weeks；2) venetoclax 200mg/d × 2 weeks 3) azacitidine 100mg/d d1-7 dicitabine combined with liposome mitoxantrone, cytarabine, and G-CSF (D-MAG) regimen 28 days per cycle ×2 cycles；
  1）dicitabine 25mg d1-3，2）liposome mitoxantrone 20mg d4，3）cytarabine 10mg/m2 Q12h d1-7 4）G-CSF 300ug d-1 until WBC > 20×109/L

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of Venetoclax Combining Chidamide and Azacitidine (VCA) Followed by D-MAG Regimen on the Treatment of Elderly Patients With Newly Diagnosed Acute Myeloid Leukemia (AML)

DETAILED DESCRIPTION:
Elderly Patients with AML have inferior outcomes due to poor physical condition, and intolerant to conventional chemotherapy. The regimen of Venetoclax and Azacitidine has been widely used in these patients and has proved to achieve higher CR rate than low intensity therapy. However, the median duration of response (DOR) of this regimen is about one year. Chidamide is a histone deacetylase (HDAC) inhibitor and preclinical data showed adding low-dose Chidamide to venetoclax could significantly promoted apoptosis of leukemia cell lines. The Venetoclax Combining Chidamide and Azacitidine (VCA) regimen was applied to one 62-year-old male patient with AML who achieved CR. Meanwhile, Liposome mitoxantrone has better safety and tolerance than mitoxantrone in elderly patients. Thus, this study is intended to use 2 cycles of VCA regimens followed by 2 cycles of D-MAG regimens, and then repeat the above four courses of treatment once to improve the median event free survival of elderly AML patients.

ELIGIBILITY:
Inclusion Criteria:

* 1) Histologically confirmed acute myeloid leukemia (non-M3). Treatment-na?ve and unable to receive standard cytarabine and anthracycline induction regimens due to age or comorbidities or patient preference.

  2) Age ≥ 60 years old, male or female, with an expected survival more than 3 months.

  3) Estimated creatinine clearance ≥ 30 mL/min. 4) AST and ALT ≤ 3.0 x ULN (unless leukemic organ involvement). Bilirubin ≤ 1.5 x ULN (unless considered due to leukemic organ involvement).

  5) ECOG ≤ 2. 6) Able to understand and voluntarily provide informed consent.

Exclusion Criteria:

* 1)Acute promyelocytic leukemia (APL) and low risk cytogenetics such as t(8;21), inv(16) or t(16;16).

  2) Active central nervous system leukemia. 3) History of myeloproliferative neoplasm (MPN) including myelofibrosis, essential thrombocythemia, polycythemia vera, chronic myeloid leukemia (CML) with or without BCR-ABL1 translocation and AML with BCR- ABL1 translocation.

  4) HIV positive patients and/or HBV or HCV active infection (documented by HBV-DNA and HCV-RNA positive test) 5) Patients suffering from chronic respiratory diseases that require continuous oxygen inhalation, or a history of obvious renal, nervous system, psychiatric, endocrine, metabolic, immune, liver, and cardiovascular diseases 6) Patients suffering from malabsorption syndrome or other conditions that exclude enteral route of administration.

  7) Patients has clinically significant QTc prolongation (>450 ms in men; >470 ms in women), ventricular tachycardia and atrial fibrillation, second-degree heart block, myocardial infarction within the year prior to enrollment, and congestive heart failure;and patients with coronary heart disease with clinical symptoms requiring drug treatment.

  8) Active, uncontrolled severe infection. 9) History of other malignancies within 2 years, except for the following: Adequately treated cervix or breast cancer in situ; Basal cell cancer or local squamous cell carcinoma of the skin; 10) White blood cell count > 25 × 10^9/L. (Hydroxyurea or leukapheresis may meet this criterion.) 11) Mental disorders that hinder research participation 12) Participants have received the following treatments: hypomethylating agents, veneclax and/or chemotherapy for myelodysplastic syndrome (MDS), solid organ transplantation.

  13) Any other circumstances that the investigator believes that the patient is not suitable to participate in this trial

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Complete remission (CR) rate | 6 months
  CR was <5% marrow blasts by morphology

SECONDARY OUTCOMES:
1 year leukemia free survival (LFS) | 1 year from treatment initiation
  Leukemia-free survival (LFS) is defined as survival without evidence of relapse from treatment initiation
1 year overall survival (OS) | 1 year from treatment initiation
  Overall survival（OS）is defined as the time from treatment initiation to death from any cause.
Adverse events | 6 months
  Adverse event is defined as any untoward medical occurrence associated with treatment
objective response rate (ORR) | 6 months
  ORR is defined as CR, CRi and PR. Partial remission (PR) is defined as a decrease of at least 50% in the percentage of blasts to 5 to 25% in the bone marrow aspirate and the normalization of blood counts.

CONTACTS AND LOCATIONS:
Overall Officials: Bing Xu, M.D., Principal Investigator — The First Affiliated Hospital of Xiamen University
Locations (1):
- Bing Xu, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: No